CLINICAL TRIAL: NCT00616980
Title: Injection of Autologous CD34-Positive Cells for Improved Symptomatic Relief and Ischemic Wound Healing in Subjects With Moderate or High-Risk Critical Limb Ischemia
Brief Title: Injection of Autologous CD34-Positive Cells for Critical Limb Ischemia
Acronym: ACT34-CLI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Losordo, Douglas, M.D. (Individual)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Director, Feinberg Cardiovascular Research Institute, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00009937/STU00001469; 11931-02 (Other: Sponsor protocol number)
Record Dates: First submitted 2008-01-24; First posted 2008-02-15 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Peripheral Artery Disease; Peripheral Vascular Disease; Critical Limb Ischemia
Keywords: PAD; PVD; CLI; Stem Cells
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose (Active Comparator)
  Interventions: Biological: CD34-positive cells
- High Dose (Active Comparator)
  Interventions: Biological: CD34-positive cells
- Saline (Placebo Comparator)
  Interventions: Biological: Saline and 5% autologous plasma

INTERVENTIONS:
Biological: CD34-positive cells
  Arms: Low Dose
Biological: CD34-positive cells
  Arms: High Dose
Biological: Saline and 5% autologous plasma
  Arms: Saline

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of intramuscular injections of adult stem cells in patients with Critical Limb Ischemia (CLI).

ELIGIBILITY:
Inclusion Criteria:

* 21-80 years of age
* moderate or high-risk Critical Limb Ischemia (Rutherford Clinical Severity Score 4 or 5)
* unsuitable for conventional revascularization

Exclusion Criteria:

* advanced CLI (Rutherford Clinical Severity Score 6) characterized by extensive tissue loss or gangrene
* advance AV block or NYHA Class III or Class IV heart failure
* myocardial infarction within 3 months of treatment
* successful coronary or lower extremity revascularization within 3 months of study enrollment
* arterial insufficiency in the lower extremity is the result of a non-atherosclerotic disorder with the exception of thromboangitis obliterans (Buerger's Disease)
* co-morbidity associated with life expectancy of less than 1 year

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-12; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Safety of Intramuscular Injection of CD34-positive cells | 6 months and 1 year
Change in Rest Pain | 6 months
Ulcer Healing | 6 months
Functional Improvement | 6 months
Limb Salvage | 6 months

SECONDARY OUTCOMES:
Disease Severity | 6 months
Assessment of Co-morbidity | 6 months

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Cardiology, PC, Birmingham, Alabama
  - Florida Research Network LLC, Gainsville, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mount Sinai School of Medicine Division of Vascular Surgery, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals of Cleveland, Case Medical Center, Cleveland, Ohio
  - University of Utah-Vascular Surgery Division, Salt Lake City, Utah
  - Swedish Medical Center, Seattle, Washington
  - Comprehensive Cardiovascular Care St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Moazzami B, Mohammadpour Z, Zabala ZE, Farokhi E, Roohi A, Dolmatova E, Moazzami K. Local intramuscular transplantation of autologous bone marrow mononuclear cells for critical lower limb ischaemia. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD008347. doi: 10.1002/14651858.CD008347.pub4. PMID 35802393
- [Derived] Losordo DW, Kibbe MR, Mendelsohn F, Marston W, Driver VR, Sharafuddin M, Teodorescu V, Wiechmann BN, Thompson C, Kraiss L, Carman T, Dohad S, Huang P, Junge CE, Story K, Weistroffer T, Thorne TM, Millay M, Runyon JP, Schainfeld R; Autologous CD34+ Cell Therapy for Critical Limb Ischemia Investigators. A randomized, controlled pilot study of autologous CD34+ cell therapy for critical limb ischemia. Circ Cardiovasc Interv. 2012 Dec;5(6):821-30. doi: 10.1161/CIRCINTERVENTIONS.112.968321. Epub 2012 Nov 27. PMID 23192920